CLINICAL TRIAL: NCT04228692
Title: Evaluation of the Benefits of Percutaneous Posterior Tibial Nerve Stimulation in Post-operative Voiding Dysfunction After Deep Endometriosis Surgery
Brief Title: Percutaneous Posterior Tibial Nerve Stimulation in Post-operative Voiding Dysfunction After Deep Endometriosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL19_0686; 2019-A02583-54 (Other: ANSM)
Record Dates: First submitted 2020-01-09; First posted 2020-01-14 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Endometriosis; Dysuria
Keywords: deep endometriosis surgery; voiding dysfunction; self-catheterization; posterior tibial nerve stimulation
MeSH Terms: conditions — Endometriosis; Dysuria

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-catheterization only (Active Comparator): Patients self-catheterized after each micturition, noting the volume of each spontaneous micturition as well as the volume obtained by subsequent self-catheterization, until self-catheterization is no longer necessary
  Interventions: Procedure: Self-catheterization only
- Posterior tibial nerve stimulation + self-catheterization (Experimental): Patients self-catheterized after each micturition, noting each volume of spontaneous micturition and each volume obtained by self-catheterization.
  Patients will have 2 sessions per day of PTN (10-20 min) until self-catheterization is no longer necessary.
  Interventions: Device: Posterior tibial nerve stimulation + self-catheterization

INTERVENTIONS:
Procedure: Self-catheterization only — Patients self-catheterized after each micturition, noting the volume of each spontaneous micturition as well as the volume obtained by subsequent self-catheterization, until self-catheterization is no longer necessary.
  Arms: Self-catheterization only
Device: Posterior tibial nerve stimulation + self-catheterization — Patients self-catheterized after each micturition, noting the volume of each spontaneous micturition as well as the volume obtained by subsequent self-catheterization, until self-catheterization is no longer necessary.
  Patients will have 2 sessions per day of PTN (10-20 min) until self-catheterization is no longer necessary.
  Arms: Posterior tibial nerve stimulation + self-catheterization

SUMMARY:
Symptomatic endometriosis can be responsible for urinary problems as well as symptoms of clinical bladder hyperactivity and/or symptoms of bladder pain before or during miction that can persist after bladder voiding. Whereas urinary problems can predate surgery due to the endometrial lesions themselves, the surgery can also have functional consequences for urinary function, specifically when there is trauma (incisions, per-operative coagulation) to the inferior hypogastric nerve fibers and/or to the hypogastric plexus.

The incidence of post-surgery urinary symptoms could be as high as 30%. The incidence of voiding problems and specifically of non-obstructive voiding dysfunction can be observed in 17,5% of cases of patients 1-month post-surgery for deep colorectal endometriosis, and persists in 4,8% of women after 12 months.

The gold standard for treatment of voiding problems consists of self-catheterization, as is the case for all non-obstructive voiding dysfunction symptoms. This procedure considerably impacts quality of life. The proper and complete voiding of the bladder remains essential in order to avoid recurring urinary tract infections and pelvic static disorder.

In the case of persistent dysuria, the use of self-catheterization is necessary in 21% of patients after surgery for deep endometriosis, for an average duration of 85 days. To date, few studies have explored the management of post-operative urinary complications after surgery for deep endometriosis. Pharmaceutical alternatives (alpha-blockers, anticholinergics, benzodiazepines) have not proven effective and sometimes cause side effects. However promising alternative treatments are being developed, specifically the neuromodulation of the sacral root. This procedure has been shown effective in the treatment of non-obstructive voiding dysfunction; however, it remains an invasive treatment that has its load of complications and undesirable side-effects. A recent study reports favorable results for the use of sacral neuromodulation in the case of persistent incomplete voiding following surgery for deep colorectal endometriosis. Some studies have also suggested that percutaneous posterior tibial nerve stimulation (PTN) could also be a treatment alternative. The advantage of this procedure is that it is non-invasive and less constraining. No study has yet evaluated whether PTN could also be used to treat patients with persistent voiding dysfunction following surgery for deep endometriosis.

Our study, conducted in the gynecologic department of Croix ROUSSE Hospital, Lyon (France), evaluates PTN as a new treatment option for post-operative voiding dysfunction in women who suffer from deep endometriosis. Our aim is to prove that the use of PTN can reduce the duration of self-catheterization by 50% when compared to self-catheterization only.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are eligible for the French public healthcare system
* Patients who have given their consent for this research

Exclusion Criteria:

* Patients with cognitive, psychiatric or motor disturbances, that do not allow for independent use of the device
* Patients who do not speak French
* Patients who have had a surgery (bladder or ureters) for endometriosis or any other reason.
* Patients who were participating in another ongoing study, or within the exclusion time stipulated by another study (at the discretion of the investigator)
* Patients unable to give their consent (protected by law: under guardianship / trusteeship)
* Patients who are taking a pharmaceutical treatment for urological problem (anticholinergics, alpha-blockers, prostaglandin)
* Pregnant or breastfeeding women
* Patients with a pacemaker
* Patients with dermatological problem in the area where the device's electrodes have to be installed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-03-11 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Reduction of 50% of total duration of self-catheterization in the self-catheterization + PTN group | From the day of surgery to the end of self-catheterization or until a maximum of 3 months
  Comparison of total numbers of days of self-catheterization between the 2 groups

SECONDARY OUTCOMES:
Number of self-catheterizations per day | From the day of surgery to the end of self-catheterization or until a maximum of 3 months
  Patients will complete a voiding calendar as long as self-catheterization is required
Post voiding residual urine volume (PVR) | From the day of surgery to the end of self-catheterization or until a maximum of 3 months
  Patients will complete a voiding calendar as long as self-catheterization is required
number of PVR> 50% of spontaneous miction | From the day of surgery to the end of self-catheterization or until a maximum of 3 months
  Patients will complete a voiding calendar as long as self-catheterization is required
side effects of PTN | From the day of surgery to the end of self-catheterization or until a maximum of 3 months
  sensation of small electrical discharges, skin reactions next to the electrodes will be notified by patients
number of sessions of PTN per week | From the day of surgery to the end of self-catheterization or until a maximum of 3 months
duration of each session of PTN | From the day of surgery to the end of self-catheterization or until a maximum of 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie WAREMBOURG, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France